CLINICAL TRIAL: NCT05720117
Title: A First-in-Human, Open-label, Multicenter, Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of PYX-201 in Participants With Advanced Solid Tumors
Brief Title: Study of PYX-201 in Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pyxis Oncology, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PYX-201-101; 2023-509687-14-00 (EU CTIS Number); 2022-002284-30 (EudraCT Number)
Record Dates: First submitted 2023-01-30; First posted 2023-02-09 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor; Advanced Solid Tumor
Keywords: Relapsed/refractory Solid Tumor; PYX-201
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1: PYX-201 Dose Escalation (Experimental): Participants will receive escalating doses of PYX-201 as an intravenous (IV) infusion to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and antitumor activity of PYX-201. Intra-participant dose escalation may be considered for participants who have adequately tolerated therapy.
  Interventions: Drug: PYX-201
- Part 2: Cohort A (Experimental): Participants with recurrent, persistent, and/or metastatic head and neck squamous cell carcinoma (HNSCC) who have received at least one but no more than two lines of prior systemic therapy, including platinum-based therapy and a programmed cell death protein 1 (PD-1) inhibitor, and participants who have received up to two lines of prior therapy that must include one prior PD-1 inhibitor and one prior epidermal growth factor receptor (EGFR)-directed treatment, will receive PYX-201 as an IV infusion at the recommended dose for Part 2.
  Interventions: Drug: PYX-201
- Part 2: Cohort B (Experimental): Participants with triple-negative breast cancer (TNBC) who have been treated with at least one but no more than two lines of prior systemic therapy will receive PYX-201 as an IV infusion at the recommended dose for Part 2.
  Interventions: Drug: PYX-201
- Part 2: Cohort C (Experimental): Participants with hormone receptor (HR)-positive (HR+)/human epidermal growth factor receptor 2 (HER2)-negative (immunohistochemistry [IHC] 0, IHC 1+, or IHC 2+/in situ hybridization [ISH]-negative) breast cancer who had progressed on cyclin-dependent kinase 4/6 (CDK-4/6) inhibitors plus endocrine therapy and one line of chemotherapy, and had received no more than three prior lines of systemic therapy, will receive PYX-201 as an IV infusion at the recommended dose for Part 2.
  Interventions: Drug: PYX-201
- Part 2: Cohort D (Experimental): Participants with various advanced solid tumor types, including non-small cell lung cancer (NSCLC), sarcomas, rare solid tumor head and neck (H&N) cancers, ovarian cancer (OVCA), cervical cancer, and endometrial cancer, will receive PYX-201 as an IV infusion at the recommended dose for Part 2.
  Interventions: Drug: PYX-201

INTERVENTIONS:
Drug: PYX-201 — IV infusion

SUMMARY:
The primary objectives of this study are to determine the recommended dose(s) of PYX-201 for participants with relapsed/refractory (R/R) solid tumors, and to determine the objective response rate (ORR) in participants treated with PYX-201 as a single agent.

ELIGIBILITY:
Inclusion

1. Histologically or cytologically confirmed solid tumors including locally advanced/metastatic NSCLC, HR+ and HER2- breast cancer, HR- and HER2-positive breast cancer, TNBC, HNSCC, ovarian cancer, thyroid cancer, pancreatic ductal adenocarcinoma (PDAC), sarcomas, hepatocellular carcinoma (HCC), kidney cancer, cervical cancer and endometrial cancer.
2. Male or non-pregnant, non-lactating female participants age ≥18 years.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 1.
4. Participant must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
5. Life expectancy of >3 months, in the opinion of the Investigator.
6. Corrected QTcF <470 msec.
7. Adequate hematologic function.
8. Adequate hepatic function.
9. Adequate renal function.
10. Adequate coagulation profile.
11. Clinical sites must conduct fresh tumor biopsy or provide participant's archived tumor tissue sample.

Exclusion

1. History of another malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin; in situ cervical carcinoma; adequately treated, noninvasive bladder cancer.
2. Known symptomatic brain metastases.
3. Significant cardiovascular disease within 6 months prior to start of study drug.
4. Evidence of an active systemic bacterial, fungal, or viral infection requiring treatment at the start of study drug.
5. Known active hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS).
6. Failure to recover to baseline severity or Grade ≤1 NCI-CTCAE v5.0 from acute non-hematologic toxicity.
7. Participants with NCI-CTCAE v5.0 Grade >1 neuropathy of any etiology.
8. Prior solid organ or bone marrow progenitor cell transplantation.
9. Prior high-dose chemotherapy requiring stem cell rescue.
10. Received systemic anticancer therapy within 28 days or within 5 half-lives (whichever is shorter) prior to the start of study drug.
11. Palliative radiation therapy within 14 days prior to the start of study drug.
12. Previously received extra domain B splice variant of fibronectin (EDB+FN) targeting treatments at any time prior to the start of PYX-201 treatment.
13. History of uncontrolled diabetes mellitus.
14. History of Stevens-Johnson syndrome or toxic epidermal necrolysis.
15. Participants with corneal epithelial disease, with the exception of mild punctate keratopathy
16. Participants with the best-corrected visual acuity in the worst-seeing eye worse than 20/100 (Snellen equivalent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants who Experience a Dose-limiting Toxicity (DLT) | Day 1 to Day 21
  DLT is defined as (1) an adverse event (AE) or abnormal laboratory value assessed as unrelated to disease, disease progression, intercurrent illness, or concomitant medications that occurs after the treatment with PYX-201 and (2) meets any of the predefined criteria outlined in the protocol.
Part 1: Number of Participants who Experience an AE | Up to approximately 3 years
  Type, incidence, seriousness, relationship to study treatment and severity of AEs, including serious AEs and AEs at Grade 3 or above, based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0. Any clinically significant changes in clinical laboratory parameters, vital signs, and electrocardiogram (ECG) parameters will be recorded as AEs.
Part 2: Objective Response Rate (ORR) | Up to approximately 2 years

SECONDARY OUTCOMES:
Part 1: Maximum Observed Concentration (Cmax) of PYX-201 Antibody-drug Conjugate, Total Antibody, Free Payload and Associated Metabolites in Serum | Day 1 up to approximately 2 years
Part 1:Time to Maximum Concentration (Tmax) of PYX-201 Antibody-drug Conjugate, Total Antibody, Free Payload and Associated Metabolites in Serum | Day 1 up to approximately 2 years
Part 1:Clearance (CL) of PYX-201 Antibody-drug Conjugate, Total Antibody, Free Payload and Associated Metabolites in Serum | Day 1 up to approximately 2 years
Part 1:Area Under the Concentration-time Curve from Time 0 to the Last Quantifiable Concentration (AUC0-t) of PYX-201 Antibody-drug Conjugate, Total Antibody, Free Payload and Associated Metabolites in Serum | Day 1 up to approximately 2 years
Part 1:Area Under the Concentration-time Curve Over the Dosing Interval (AUCtau) of PYX-201 Antibody-drug Conjugate, Total Antibody, Free Payload and Associated Metabolites in Serum | Day 1 up to approximately 2 years
Part 1:Area Under the Concentration-time Curve from Time 0 Extrapolated to Infinity (AUC0-inf) of PYX-201 Antibody-drug Conjugate, Total Antibody, Free Payload and Associated Metabolites in Serum | Day 1 up to approximately 2 years
Part 1:Half-life (t½) of PYX-201 Antibody-drug Conjugate, Total Antibody, Free Payload and Associated Metabolites in Serum | Day 1 up to approximately 2 years
Part 1: ORR | Up to approximately 3 years
Part 1:Duration of Response (DOR) | Up to approximately 3 years
Part 1:Progression-free Survival (PFS) | Up to approximately 3 years
Part 1:Disease Control Rate (DCR) | Up to approximately 3 years
Part 1:Time to Response (TTR) | Up to approximately 3 years
Part 1:Overall Survival (OS) | Up to approximately 3 years
Part 1:Number of Participants With Anti-drug Antibodies to PYX-201 | Up to approximately 2 years
Part 2: DOR | Up to approximately 2 years
Part 2: Clinical Benefit Rate | Up to approximately 2 years
Part 2: Median Progression-free Survival (mPFS) | Up to approximately 4 years
Part 2: DCR | Up to approximately 2 years
Part 2: TTR | Up to approximately 2 years
Part 2: Median Overall Survival (mOS) | Up to approximately 4 years
Part 2: Cmax of PYX-201 | Up to approximately 2 years
Part 2: Tmax of PYX-201 | Up to approximately 2 years
Part 2: Trough Concentration of PYX-201 | Up to approximately 2 years
Part 2: Number of Participants who Experience an AE | Up to approximately 2 years
  Type, incidence, seriousness, relationship to study treatment and severity of AEs, including serious AEs and AEs at Grade 3 or above, based on NCI-CTCAE Version 5.0. Any clinically significant changes in clinical laboratory parameters, vital signs, and ECG parameters will be recorded as AEs.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (10):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - SCRI - HealthOne Denver, Denver, Colorado
  - SCRI - Florida Cancer Specialists, Sarasota, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Rhode Island Hospital, Providence, Rhode Island
  - NEXT Dallas, Dallas, Texas
  - NEXT San Antonio, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia
- Belgium (4):
  - Institut Jules Bordet, Brussels, Brussels Capital
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
- Spain (5):
  - Hospital Universitari Vall d'Hebrón, Barcelona, Barcelona
  - START Madrid - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia, València
- Sarah Cannon Research Institute London, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No